CLINICAL TRIAL: NCT04329728
Title: An Open Label, Phase 1/2 Study Evaluating Immunomodulatory AVM0703 in Patients With Lymphoid Malignancies (OPAL Study)
Brief Title: The OPAL Study: AVM0703 for Treatment of Lymphoid Malignancies
Acronym: OPAL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AVM Biotechnology Inc (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVM0703-001
Record Dates: First submitted 2020-03-13; First posted 2020-04-01 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Lymphoid Malignancies
Keywords: Diffuse large B-cell lymphoma (DLBCL); B-cell lymphoma; Mantle cell lymphoma (MCL); Primary mediastinal large B-cell Lymphoma; Primary DLBCL of the central nervous system (CNS); Burkitt or Burkitt-like lymphoma/leukemia; Chronic lymphocytic leukemia (CLL); Small lymphocytic leukemia (SLL); B-cell leukemia/lymphoma; T-cell leukemia/lymphoma; Acute leukemias of ambiguous lineage; Natural Killer (NK) cell lymphoblastic leukemia/lymphoma; Advanced or Aggressive lymphoma/lymphoproliferative disease; Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, B-Cell; Lymphoma, Mantle-Cell; Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell; Lymphoma; Leukemia, T-Cell; Leukemia, Biphenotypic, Acute; Lymphoproliferative Disorders; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- DLBCL and high-grade B-cell lymphoma (Experimental): Diffuse Large Cell B-Lymphoma High-grade B-cell Lymphoma
  Interventions: Drug: AVM0703
- MCL (Chronic Lymphoid Leukemia) (Experimental): Chronic Lymphoid Leukemia
  Interventions: Drug: AVM0703
- Primary Mediastinal Large B-cell lymphoma (Experimental): Primary mediastinal large B-cell lymphoma
  Interventions: Drug: AVM0703
- Burkitt or Burkitt-like lymphoma/leukemia (Experimental): Burkitt or Burkitt-like lymphoma/leukemia
  Interventions: Drug: AVM0703
- CLL/SLL (Experimental): Chronic Lymphocytic Leukemia Small Lymphocytic Lymphoma
  Interventions: Drug: AVM0703
- B- or T-ALL (Experimental): B-lymphoblastic leukemia/lymphoma, T-lymphoblastic leukemia/lymphoma, acute leukemia/lymphoma, acute leukemias of ambiguous lineage, or natural killer (NK) cell lymphoblastic leukemia/lymphoma
  Interventions: Drug: AVM0703

INTERVENTIONS:
Drug: AVM0703 — Intravenous infusion over ~1 hours
  Other Names: Supra-Pharmacologic Dexamethasone Phosphate

SUMMARY:
This is an open-label, Phase 1/2 study designed to characterize the safety, tolerability, Pharmacokinetics(PK), and preliminary antitumor activity of AVM0703 administered as a single intravenous (IV) infusion to patients with lymphoid malignancies.

DETAILED DESCRIPTION:
Phase 2 For Phase 2, one or more patient cohort(s) will receive repeat RP2D infusions in 21 day intervals until intolerance, unacceptable toxicity or disease progression, to determine the number of repeat infusions that are safe, effective and tolerable in this patient population. PK assessments will be made at sites participating in both Phase 1 and Phase 2 after each repeat infusion for the first 6 patients enrolled into each repeat dosing cohort. Full PK assessments will be made as per Phase 1 after the 1st (first) and 6th (sixth) repeat infusions, while for the second to fifth doses (2nd to 5th) PK assessments will be made pre-infusion, at end of infusion, 15 minutes and 48 hours after end of infusion. At least 6 patients will be enrolled in each RP2D repeat dosing cohort. The DSMC will monitor unacceptable toxicities during Phase 2 and halting/stopping criteria are outlined in Table 6. After 6 patients, who have had PK assessments, have reached intolerance, unacceptable toxicity, or disease progression, or they have received 6 infusions without intolerance, unacceptable toxicity, or disease progression, the Data Safety Monitoring Committee will review an integrated interim analysis of all available PK, PD, efficacy, safety and tolerability data and determine whether repeat dosing should continue or be limited to a certain number of infusions. Ongoing DSMC review will occur at least every 6 months. Based on integrated analysis, including dose-response and exposure-response, the DSMC will determine the optimal dose and dosing schedule for repeat dosing with AVM0703.

For Phase 2, RP2D cohorts will be included that do not require repeat 21 day interval dosing for patients who cannot comply with the visit schedule for repeat dosing. These patients can be retreated according to section 5.5.3.2.

An 18 mg/kg dose (expressed as dexamethasone phosphate) has been approved by the SRC for an RP2D. The 21 mg/kg dose-escalation cohort remains open for dose-escalation enrollment. For sites participating in both Phase 1 and Phase 2, patients will be enrolled into the 21 mg/kg dose-cohort unless i) no slot is available, ii) the patient cannot logistically comply with the PK blood draw requirements, iii) the cohort has been fully enrolled, or iv) the patient is enrolled into a Phase 2 repeat dosing RP2D cohort.

For prophylaxis against dexamethasone-induced CNS side effects, hydrocortisone will be dosed orally for 5 days starting on the day of dexamethasone infusion. Hydrocortisone will be divided into 3 daily doses starting in the morning and spaced 6 to 8 hours apart using the following dosing schedule each day: for pediatric and adolescent patients at 5 mg/m2 (morning dose), 3 mg/m2 (mid day dose), and 2 mg/m2 dose (evening dose); and for adult patients at 10 mg/m2 (morning dose), 5 mg/m2 (mid-day dose), and 5 mg/m2 dose (evening dose), the last dose administered at hour of sleep.

* Prophylaxis for GI bleeding: Administer a proton pump inhibitor or H2 blocker starting at least 1 day prior to and for approximately 4 weeks after AVM0703 administration, as per institutional guidelines.
* Prophylaxis for TLS: All patients should be assessed for risk of TLS. Patients at high risk for TLS are defined as patients with ALC >25 × 109/L and/or who have a lymph node >10 cm. For patients at high risk of TLS, recommended prophylaxis is oral and IV hydration and anti hyperuricemic therapy (eg, allopurinol or rasburicase) starting at 2 days before AVM0703 administration.
* Prophylaxis for patients not deemed high risk for TLS will be at the discretion of the Investigator.
* Monitoring TLS: High-risk patients should have TLS labs (eg, potassium, phosphorus, calcium, uric acid, and creatinine) obtained predose, and 4 and 8 hours post-infusion of AVM0703 on Day 0.

The Phase 2 portion of the study will include patients with malignancies that are potentially responsive to AVM0703, such as DLBCL (including DLBCL arising from follicular lymphoma and primary DLBCL of the CNS), high-grade B-cell lymphoma or Burkitt lymphoma, Chronic lymphocytic leukemia (CLL)/ SLL, T-cell lymphoma, or Acute lymphoblastic leukemia (ALL). Up to approximately 18 patients will be enrolled into each of the selected tumor types at the MTD/RP2D defined in the Phase 1 portion of the study.

For patients not enrolled into 21 day repeat dosing cohorts, upon disease relapse, patients may be retreated at a dose previously shown to be safe. If a patient must be given additional anticancer therapy before Day 28, disease assessment should be performed before they receive any other therapy. Patients who go on to receive additional anticancer therapy will be followed for survival at 3, 6, and 12 months post-infusion, and yearly thereafter until death, withdrawal of consent/assent, or study closure. Survival information can be obtained via public records, telephone calls, and/or medical records. Any subsequent anticancer therapy that the patients receive will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥12 years and weight ≥40 kg;

  2. Histologically confirmed diagnosis per 2016 World Health Organization (WHO) classification of lymphoid neoplasms160 and per the 2016 WHO classification of acute leukemia161 of the following indications:
  * DLBCL, including arising from follicular lymphoma;
  * High-grade B-cell lymphoma;
  * MCL;
  * Primary mediastinal large B-cell lymphoma;
  * Primary DLBCL of the CNS;
  * Burkitt or Burkitt-like lymphoma/leukemia;
  * CLL/SLL; or
  * B-lymphoblastic leukemia/lymphoma, T-lymphoblastic leukemia/lymphoma, acute leukemia/lymphoma, acute leukemias of ambiguous lineage, or NK cell lymphoblastic leukemia/lymphoma;

    3. Patients must have relapsed or refractory (R/R) disease with prior therapies defined below:
  * DLBCL and high-grade B-cell lymphoma:

    e) R/R after autologous hematopoietic cell transplant (HCT); or f) R/R after chimeric antigen receptor T-cell (CAR T) therapy; or g) Patients not eligible for autologous HCT or CAR T therapy; or h) R/R after ≥2 lines of therapy including anti-CD20 antibody and failed, intolerant or ineligible for polatuzamab vedotin, or for whom no standard therapy is available.
  * MCL:

    c) R/R after autologous HCT; or d) Patients not eligible for autologous HCT must have failed acalabrutinib or be R/R after ≥2 lines of therapy including at least 1 of the following: a Bruton's tyrosine kinase (BTK) inhibitor, bortezomib, or lenalidomide; or for whom no standard therapy is available;
  * Primary mediastinal large B-cell lymphoma: R/R after ≥1 line of therapy and are not eligible for or have recurred after autologous HCT or CAR T cell therapy, or for whom no standard therapy is available;
  * Primary DLBCL of the CNS: R/R after ≥1 line of therapy including methotrexate (unless intolerant to methotrexate) and are not eligible for or have recurred after autologous HCT or CAR T cell therapy, or for whom no standard therapy is available;
  * Burkitt or Burkitt-like lymphoma/leukemia: R/R after ≥1 line of therapy including methotrexate (unless intolerant to methotrexate) and are not eligible for or have recurred after autologous HCT or CAR T cell therapy, or for whom no standard therapy is available;
  * CLL/SLL: patients who have active disease requiring treatment and who are deemed at high-risk for disease progression by the investigator or have high risk features per the iwCLL criteria, such as primary resistance to first-line chemo(immune)therapy, or progression of disease <3 years after fludarabine-based chemo(immune)therapy, or leukemia cells with del(17p)/TP53 mutation, must be:

    d) R/R after autologous or allogeneic HCT; or e) Patients not eligible for HCT; or f) R/R after ≥2 lines of therapy including at least 1 of the following: a BTK inhibitor, venetoclax, idelalisib, or duvelisib, or for whom no standard therapy is available;
  * Acute lymphoblastic leukemia (ALL):

    c) R/R after allogeneic HCT and for whom no standard therapy is available; or d) Patients not eligible for allogeneic HCT must be R/R according to the following disease specific specifications:
  * B-cell lymphoblastic leukemia/lymphoma: ≥2 lines of therapy including approved CAR T cell therapies, inotuzumab ozogamicin, or blinatumomab, or for whom no standard therapy is available;
  * T-cell lymphoblastic leukemia/lymphoma: ≥2 lines of therapy including nelarabine, or for whom no standard therapy is available;
  * NK cell leukemia/lymphoma: ≥1 line of therapy or for whom no standard therapy is available;
  * All other diagnoses: R/R after autologous or allogeneic HCT; or R/R after at least one line of therapy, or for whom no standard therapy is available.

    4. Lansky (12 to 15 years of age) (Appendix G) or Karnofsky (≥16 years of age) (Appendix H) performance status ≥50;

    5. Screening laboratory values that meet all of the following criteria:
  * Absolute neutrophil count ≥0.05 × 109/L;
  * Platelet count ≥25 × 109/L;
  * Hemoglobin ≥6.5 g/dL;
  * • Aspartate aminotransferase or alanine aminotransferase ≥2.5 × ULN, unless due to the disease;
  * Total bilirubin <1.5 × ULN (if secondary to Gilbert's syndrome, <3 × ULN is permitted), unless due to the disease; and
  * Glomerular filtration rate ≥30 mL/min ; except for patients on metformin at baseline GFR must be ≥45 mL/min; GFR can be calculated by the Cockcroft-Gault formula Appendix C);

    6. Minimum level of pulmonary reserve defined as <Grade 2 dyspnea and pulse oximetry ≥92% on room air;

    7. Females of childbearing potential must have a negative serum pregnancy test at screening. Females of childbearing potential and nonsterile males must agree to use medically effective methods of contraception from the time of informed consent/assent through 1 month after study drug infusion, which must, at a minimum, include a barrier method; and

    8. The ability to understand and willingness to sign a written informed consent form (ICF) and the ability to adhere to the study schedule and prohibitions. Patients under the age of 18 years (or other age as defined by regional law or regulation) must be willing and able to provide written assent and have a parent(s) or guardian(s) willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to performance of any study-related procedure.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from participation in the study for Phase 2:

  1. History of another malignancy, except for the following:

     * Adequately treated local basal cell or squamous cell carcinoma of the skin;
     * Adequately treated carcinoma in situ without evidence of disease;
     * Adequately treated papillary, noninvasive bladder cancer; or
     * Other cancer that has been in complete remission for ≥2 years. Patients with low-grade prostate cancer, on active surveillance, and not expected to clinically progress over 2 years are allowed;
  2. Significant cardiovascular disease (e.g., myocardial infarction, arterial thromboembolism, cerebrovascular thromboembolism) within 3 months prior to the start of AVM0703 administration, angina requiring therapy, symptomatic peripheral vascular disease, New York Heart Association Class III or IV congestive heart failure, left ventricular ejection fraction <30%, left ventricular fractional shortening <20%, or uncontrolled ≥Grade 3 hypertension (diastolic blood pressure >100 mmHg or systolic blood pressure >150 mmHg) despite antihypertensive therapy for patients ≥18 years of age, or uncontrolled stage 2 hypertension (diastolic blood pressure >90 mmHg or systolic blood pressure >140 mmHg) despite antihypertensive therapy for patients ≥12 years of age;
  3. Significant screening electrocardiogram (ECG) abnormalities, including unstable cardiac arrhythmia requiring medication, atrial fibrillation/flutter, second degree atrioventricular (AV) block type 2, third-degree AV block, ≥Grade 2 bradycardia, or heart rate corrected QT interval using Fridericia's formula >480 msec;
  4. Known gastric or duodenal ulcer;
  5. Uncontrolled type 1 or type 2 diabetes;
  6. Known hypersensitivity or allergy to the study drug or any of its excipients;
  7. Untreated ongoing bacterial, fungal, or viral infection (including upper respiratory tract infections) at the start of AVM0703 administration, including the following:

     * Positive hepatitis B surface antigen and/or hepatitis B core antibody test plus a positive hepatitis B polymerase chain reaction (PCR) assay. Patients with a negative PCR assay are permitted with appropriate antiviral prophylaxis;
     * Positive hepatitis C virus antibody (HCV Ab) test. Patients with a positive HCV Ab test are eligible if they are negative for hepatitis C virus by PCR;
     * Positive human immunodeficiency virus (HIV) antibody test with detectable HIV load by PCR, or the patient is not able to tolerate antiretroviral therapy; or
     * Positive tuberculosis test during screening; test must be positive and not indeterminate due to anergy; if the result is indeterminate due to anergy the patient must not have a history of recent exposure to tuberculosis. Patients in Phase 2 repeat dosing cohorts should not travel to any destination where they might be exposed to tuberculosis during their entire treatment period with AVM0703.
  8. Received live vaccination within 8 weeks of screening;
  9. Pregnant or breastfeeding;
  10. Concurrent participation in another therapeutic clinical study (except AVM0703-001); or
  11. Uncontrolled bipolar disorder or schizophrenia. Patients with a diagnosis, past or current, of bipolar disorder or schizophrenia or having a history of severe depression or substance abuse must be prophylactically treated with circadian physiologic hydrocortisone per section 5.5.3.3 CNS prophylaxis, without exception.

Ages: 12 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2020-11-06 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: incidence of Adverse events | Year One
  The primary endpoint for the Phase 1 portion of the study is the incidence of Adverse events (AEs), including DLTs.

SECONDARY OUTCOMES:
Phase 2: ORR | Year Two
  ORR (CR plus partial response [PR]) at 28 days post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Budde, MD, Principal Investigator — City of Hope Medical Center; Gary Schiller, MD, Principal Investigator — University of California, Los Angeles; Tamra Slone, MD, Principal Investigator — U Texas SouthWestern; Don Stevens, MD, Principal Investigator — Norton Cancer Institute; Lasika Seneviratne, MD, Principal Investigator — Los Angeles Cancer Network; Pamela Miel, MD, Principal Investigator — Innovative Clinical Research Institute; Stefano Tarantolo, MD, Principal Investigator — Nebraska Cancer Specialists; Daniel Kerr, MD, Principal Investigator — ASCLEPES Research Centers; Nashat Gabrail, MD, Principal Investigator — Gabrail Cancer Center Research; Paul Rubinstein, MD, Principal Investigator — University of Illinois at Chicago; Salil Goorha, MD, Principal Investigator — Memphis Baptist Cancer Center
Locations (11):
- United States (11):
  - City of Hope, Duarte, California
  - Los Angeles Cancer Network, Los Angeles, California
  - UCLA Medical Center of Hematology/Oncology, Los Angeles, California
  - Innovative Clinical Research Institute, Whittier, California
  - ASCLEPES Research Centers, Weeki Wachee, Florida
  - University of Illinois at Chicago Cancer Center, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Gabrail Cancer Center Research,, Canton, Ohio
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - University of Texas(UT) Southwestern-Children's Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Published Abstract — https://www.alliedacademies.org/proceedings/a-novel-lymphoablation-preconditioning-agent-avm0703-via-receptor-mediated-induction-of-apoptosis-to-reduce-patient-toxi-4764.html — https://www.alliedacademies.org/proceedings/a-novel-lymphoablation-preconditioning-agent-avm0703-via-receptor-mediated-induction-of-apoptosis-to-reduce-patient-toxi-4764.html

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT04329728/Prot_SAP_000.pdf